CLINICAL TRIAL: NCT05789836
Title: The Effect Of Participation in Care Of Mothers With Newborn Baby in Surgical Intensive Care On Mother's Self-Confidence And Mother-Infant Attachment
Brief Title: The Effect of Partıcıpatıon in Care of Mothers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Mukaddes Demir Acar, Assist. Prof. Dr., Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: TOGUMDEMIRACAR
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Newborn; Attachment; Self Confidence; Nursing Caries
MeSH Terms: interventions — Nursing Care

STUDY DESIGN:
Intervention Model Description: This research was planned as a single group pretest-posttest quasi-experimental.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Experimental): This research was planned as a single group pretest-posttest quasi-experimental.
  Interventions: Other: Nursing care

INTERVENTIONS:
Other: Nursing care — Involving the mother in nursing care

SUMMARY:
The aim of the study is to examine the effect of including mothers with newborn babies in surgical intensive care units during the nursing care process on mother's self-confidence and mother-infant attachment.

DETAILED DESCRIPTION:
Population and Sample of the Research

The population of the study consists of mothers who were hospitalized with their babies in the surgical intensive care unit in a children's hospital in Ankara (Turkiye). It is planned that the mothers who were hospitalized with their babies in the surgical intensive care unit for a period of 6 months between the dates of the study and who met the criteria for inclusion in the study constitute the sample of the study.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient treatment of the baby in the surgical neonatal intensive care unit without the mother's presence since birth
* The mother stays with the baby for at least 4 days in the post-operative period
* The mother does not have any communication and language problems
* The mother's willingness to participate in the research

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Mother
Enrollment: 30 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Taylor Mother-Infant Attachment Scale | 6 month
  The answers consisting of four options are scored between 0-3, the lowest score that can be obtained from the scale is 0 and the highest score is 24.
Pharis Self-Confidence Scale | 6 month
  The Pharis Self-Confidence Scale, a 13-item, five-point measurement tool, measures a parent's feelings of self-confidence about daily baby care. Each infant care item is rated from 1 (not at all) to 5 (completely). High total score results indicate high self-confidence in babysitting.
Care Participation Assessment Scale | 6 month
  Care practices of mothers are evaluated as Yes-No and scored as 1-0. Although the maximum score that can be obtained from the scale is 19, an increase in the score means that participation in care has dropped.

CONTACTS AND LOCATIONS:
Overall Officials: Mukaddes Demir Acar, Study Chair — Tokat Gaziosmanpasa University
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Karakulak HA, Alparslan, Ö. Anne-bebek Bağlanma Ölçeğinin Türk Toplumuna Uyarlanması: Aydın Örneği. Çağdaş Tıp Dergisi. 2016; 6(3), 188-199.
- [Result] Karaçam Z, Çakmak E, Yenidoğan Yoğun Bakım Ünitesinde Bebeği Yatan Anneler İçin Bakıma Katılımı Değerlendirme Ölçeği: Ölçek Geliştirme, Geçerlilik ve Güvenilirliği. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi. 2018; 21(2), 69-78.